CLINICAL TRIAL: NCT06446609
Title: Understanding the Natural History and Impact of Itching (Pruritus) in Patients With Drug-induced Liver Injury (DILI)
Brief Title: Drug-induced Liver Injury: Itching Study
Status: Recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Ipsen (Industry); National Institute for Health Research, United Kingdom (Other Government); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23056
Record Dates: First submitted 2024-05-15; First posted 2024-06-06 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Drug Induced Liver Injury; Pruritus
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Pruritus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Idiosyncratic drug-induced liver injury (DILI) is an unpredictable adverse hepatic reaction to a medication used in its therapeutic dose. DILI is the second most common cause of itching in adult Hepatology after biliary obstruction. In particular cholestatic or mixed pattern types of DILI (in which bile flow from the liver is impaired) are associated with long-lasting effects as well as reduced quality of life. There is therefore an urgent need to determine the incidence and natural history of itching in DILI and establish a network of centres that will form a basis for a clinical trial to investigate a novel intervention to treat these.

DETAILED DESCRIPTION:
In Idiosyncratic drug-induced liver injury (DILI), the adverse effect is unexpected from the known pharmacological action of the agent. The incidence of DILI is estimated as between 14-19 per 100,000 inhabitants; a population-based study in Europe reported the annual incidence as 19.1 per 100,000. Despite its rarity, idiosyncratic DILI accounts for 7-15% of the cases of acute liver failure in Europe, although many cases resolve quickly. DILI is the most frequent reason for the market withdrawal of an approved drug. In addition, DILI occurs in association with many drugs and shows heterogeneity. There are no markers that can effectively pre-empt and prevent DILI or monitor the severity and course of the adverse event. It is also emerging that immunotherapy regimens devised for cancer treatment are associated with increased risk of DILI development.

Further characterisation and understanding of this is urgently needed to distinguish from other causes and develop more effective treatments. Age, smoking, metabolic syndrome, co-morbidity and other yet unidentified factors may generate an environment of oxidative stress that contributes to DILI. Therefore, 'in-depth phenotyping' is needed to develop a refined understanding of drug-related factors, host genetic and environmental risk factors linked to disease characteristics that would enable us to pre-empt and treat DILI. Further work is also needed to identify patients who may benefit from new treatments becoming available, so identification and analysis of certain sub-groups is of value.

Based on the pattern of liver biochemistry at the time of initial presentation, DILI is classified as cholestatic, hepatocellular or mixed type. Pruritus (itching) occurs in a proportion of patients with cholestatic and mixed pattern of DILI. Most DILI manifestations resolve within 3 months following the prompt withdrawal of the causative medication, but symptoms persist for 6 months in 18.8% and for 1 year in 12.4%; persistence of symptoms are more common in cholestatic pattern of DILI. Those with persistent DILI have significantly lower SF-36 quality of life scores at baseline and during follow-up.

Research is needed to identify patients who may benefit from new treatments becoming available, so identification and analysis of certain sub-groups is of value. DILI is the second most common cause of itching in adult Hepatology, after biliary obstruction. Cholestatic or mixed pattern of DILI is associated with chronicity as well as reduced quality of life.

There is currently limited data available on the incidence and impact of pruritus in DILI. Although therapeutics targeting bile acid pathways have been deployed to tackle cholestatic pruritus in primary biliary cholangitis (PBC), their application in cholestatic DILI requires investigation. Further, there is now also effective treatment that have been licensed to improve quality of life of patients with itching as well as potentially improving natural history of cholestatic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 (no upper age limit) and able to give informed written consent
* Exposure to potential causal agent and diagnosed with suspected acute DILI defined as meeting one of the following analytical thresholds at enrolment (visit 1):

  * alanine transaminase (ALT) ≥5 times upper limit of normal (ULN) or
  * alkaline phosphatase ≥2 times ULN or
  * ALT ≥3 times ULN plus total bilirubin >2 times ULN

Results from clinical test samples collected within 36h of visit will be acceptable (as DILI is an acute event, patients are expected to recover or deteriorate quickly so enrolment aligned with diagnostic tests is necessary).

Exclusion Criteria:

* Patients with comorbidities of eczema and urticaria associated with pruritus
* Patients with existing diagnosis of blood-borne viral hepatitis infection (Hepatitis B/C/E)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited are those who meet the criteria for DILI, as defined by Aithal et al. (2011) and endorsed by the EASL DILI Guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of pruritus (itching) in patients with DILI | 2 years
  To determine the number of participants who have diagnosis of DILI who report pruritus (itching) compared to the number with other acute non-DILI conditions (e.g. autoimmune hepatitis/viral hepatitis) who report itching within a cohort of patients presenting with acute liver injury.

SECONDARY OUTCOMES:
Duration of itching (pruritus) in patients who present with acute liver injury | 4 years
  To determine the duration and re-occurrence of pruritus (itching) symptoms in patients who are diagnosed with DILI and in those with other acute non-DILI conditions. This will entail a repeated questionnaire at study visits and assessment of medical records to report a timescale of symptoms (weeks).
Severity of itching (pruritus) in patients who present with acute liver injury | 4 years
  To determine the severity of pruritus (itching) symptoms in patients who are diagnosed with DILI and in those with other acute non-DILI conditions. This will entail a repeated questionnaire at study visits to establish the level of itching.
Genetic variants associated with itching (pruritus) in patients who present with acute liver injury | 2.5 years
  To determine whether any genetic variants of a 77 gene liver cholestasis panel (including causal variants of progressive familial intrahepatic cholestasis (PFIC)) are associated with pruritus in acute liver injury patients. The study will report presence or absence of genetic markers
Health status reported by patients who present with acute liver injury | 4 years
  To determine the health status reported by patients who are diagnosed with DILI and in those with other acute non-DILI conditions. This will entail a repeated Short Form 36 Health Survey Questionnaire (SF-36) questionnaire at study visits giving a score ranging from 0 to 100. Higher scores indicate better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

REFERENCES:
- [Background] Aithal GP, Watkins PB, Andrade RJ, Larrey D, Molokhia M, Takikawa H, Hunt CM, Wilke RA, Avigan M, Kaplowitz N, Bjornsson E, Daly AK. Case definition and phenotype standardization in drug-induced liver injury. Clin Pharmacol Ther. 2011 Jun;89(6):806-15. doi: 10.1038/clpt.2011.58. Epub 2011 May 4. PMID 21544079
- [Background] Andrade RJ, Chalasani N, Bjornsson ES, Suzuki A, Kullak-Ublick GA, Watkins PB, Devarbhavi H, Merz M, Lucena MI, Kaplowitz N, Aithal GP. Drug-induced liver injury. Nat Rev Dis Primers. 2019 Aug 22;5(1):58. doi: 10.1038/s41572-019-0105-0. PMID 31439850
- [Background] Bjornsson ES, Bergmann OM, Bjornsson HK, Kvaran RB, Olafsson S. Incidence, presentation, and outcomes in patients with drug-induced liver injury in the general population of Iceland. Gastroenterology. 2013 Jun;144(7):1419-25, 1425.e1-3; quiz e19-20. doi: 10.1053/j.gastro.2013.02.006. Epub 2013 Feb 16. PMID 23419359
- [Background] Bjornsson ES, Stephens C, Atallah E, Robles-Diaz M, Alvarez-Alvarez I, Gerbes A, Weber S, Stirnimann G, Kullak-Ublick G, Cortez-Pinto H, Grove JI, Lucena MI, Andrade RJ, Aithal GP. A new framework for advancing in drug-induced liver injury research. The Prospective European DILI Registry. Liver Int. 2023 Jan;43(1):115-126. doi: 10.1111/liv.15378. Epub 2022 Aug 15. PMID 35899490
- [Background] Chen HL, Li HY, Wu JF, Wu SH, Chen HL, Yang YH, Hsu YH, Liou BY, Chang MH, Ni YH. Panel-Based Next-Generation Sequencing for the Diagnosis of Cholestatic Genetic Liver Diseases: Clinical Utility and Challenges. J Pediatr. 2019 Feb;205:153-159.e6. doi: 10.1016/j.jpeds.2018.09.028. Epub 2018 Oct 23. PMID 30366773
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Drug-induced liver injury. J Hepatol. 2019 Jun;70(6):1222-1261. doi: 10.1016/j.jhep.2019.02.014. Epub 2019 Mar 27. PMID 30926241
- [Background] Fontana RJ, Hayashi PH, Barnhart H, Kleiner DE, Reddy KR, Chalasani N, Lee WM, Stolz A, Phillips T, Serrano J, Watkins PB; DILIN Investigators. Persistent liver biochemistry abnormalities are more common in older patients and those with cholestatic drug induced liver injury. Am J Gastroenterol. 2015 Oct;110(10):1450-9. doi: 10.1038/ajg.2015.283. Epub 2015 Sep 8. PMID 26346867
- See also: odevixibat description — https://www.ema.europa.eu/en/documents/product-information/bylvay-epar-product-information_en.pdf